CLINICAL TRIAL: NCT01395485
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 827 in Adolescent (12 to <18 Years) and Adult Subjects With Intermittent or Mild to Moderate Persistent Asthma
Brief Title: Safety, Tolerability, and Pharmacokinetics of AMG 827 in Adolescents With Asthma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study had been cancelled and replaced with protocol 20130250.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20101281
Record Dates: First submitted 2011-05-05; First posted 2011-07-15 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Asthma
Keywords: Amgen; Adolescent; Single Dose; Safety; Pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Cohort 2 (Experimental): Adolescents - Ages 13 to <17
  Interventions: Drug: AMG 827 or Placebo
- Cohort 1 (Experimental): Adolescents - Ages 12 to <13
  Interventions: Drug: AMG 827 or Placebo
- Cohort 4 (Experimental): Adults - Ages 18 to <=50
  Interventions: Drug: AMG 827 or Placebo
- Cohort 3 (Experimental): Adolescents - Ages 17 to <18
  Interventions: Drug: AMG 827 or Placebo

INTERVENTIONS:
Drug: AMG 827 or Placebo — A single dose of AMG 827 or matching placebo is to be administered subcutaneously (SC).

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics in adolescent and adult subjects with intermittent or mild to moderate persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects 12 to < 18 years of age at the time of randomization
* Male and/or female subjects between 18 and 50 years of age (inclusive) at the time of randomization
* Body weight ≥ 36 kg at screening
* Intermittent or mild to moderate persistent asthma for at least the past 3 months prior to study enrollment (as defined by the 2004 Global Initiative for Asthma [GINA] guidelines.

Exclusion Criteria:

* Experienced an asthma exacerbation (defined as a disease episode resulting in treatment in an emergency room or urgent care facility, or an episode treated with oral corticosteroids) during the 3 months prior to study enrollment.
* Hospitalized for asthma during the 6 months prior to study enrollment; or ever intubated for the treatment of asthma.
* Use of oral corticosteroids within 3 months prior to study enrollment.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment-emergent adverse events, safety and laboratory assessments in adolescent subjects with intermittent or mild to moderate asthma as a measure of safety and tolerability | Participants will be followed for the duration of the study, an expected average of 5 weeks

SECONDARY OUTCOMES:
Area under the AMG 827 concentration versus time curve (AUC) for times 0 to infinity (AUC 0-inf) and 0 to last sampling time point (AUC 0-tlast), peak plasma concentration (Cmax) and Time to peak plasma concentration (tmax) will be determined for AMG 827 | Intermittantly throughout the duration of the study, an expected average of 5 weeks
Evaluation of treatment-emergent adverse events, safety and laboratory assessments in adult subjects with intermittent or mild to moderate asthma as a measure of safety and tolerability | Intermittantly throughout the duration of the study, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com